CLINICAL TRIAL: NCT05960968
Title: Gender Specific Registry in Subjects Hospitalized With Heart Failure in Santiago( GENESIS Registry): Pilot Heart Failure Registry Looking for Sex Analysis
Brief Title: Gender Specific Registry in Subjects Hospitalized With Heart Failure in Santiago
Acronym: GENESIS
Status: Recruiting | Type: Observational
Sponsor: Fundacion de la Sociedad Chilena de Cardiologia y Cirugia Cardiovascular (Other)
Collaborators: Hospital Dipreca (Other); Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Other Study IDs: FSoChiCar-HF01
Record Dates: First submitted 2023-06-18; First posted 2023-07-27 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure
Keywords: Heart Failure,; Gender; Women; Epidemiology
MeSH Terms: conditions — Heart Failure; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational registry, which main purpose is to assess sex-related differences in heart failure (HF) presentation, management, and prognosis in patients admitted to a hospital with a certain diagnosis of HF. The diagnosis will be based on European Society of Cardiology (ESC) definition of HF ( clinical syndrome characterized by symptoms and/or signs caused by a cardiac abnormality, that results in elevated intracardiac pressure and/or inadequate output at rest or exercise ). The sample will be obtained prospectively by recruitment of patients of two hospitals of Santiago de Chile.

DETAILED DESCRIPTION:
-Methods Study design and participants

Observational and prospective registry led by the Chilean Society of Cardiology and Cardiac Surgery Foundation (Fundación SOCHICAR), that will be held at hospitals of different communes in urban Santiago. This project will incorporate two hospitals in a period of one year.

The hospital selection will be based on the purpose of having the most clinical information of the patient regarding his/her cardiac condition. Both participating centers must have coronary units, cardiac surgery, and interventional cardiology. Also, both hospitals must have medical teams with expertise in cardiac imaging, and have access to a local laboratory that performs biomarkers (i.e. NT-terminal pro-brain natriuretic peptide (NTpro-BNP), usTroponin).

The registry consists of a descriptive cross-sectional survey. Thereby, this study is a one-time assessment, with no visit schedule.

Ethics consideration The registry must be approved by the Ethics committee of each clinical center, or in case of not having one, by the Metropolitan Region Ethics Committee respective of each area. Each patient must be informed about the study's rationale and his/ her potential willingness of participation. Written informed consent will be obtained from all participants before data collection.

Study population: approximately 500 patients hospitalized in the two recruiting centers during one year who comply with all the eligible criteria and without exclusion criteria.

-Data source Data will be obtained from the medical files, and will be collected prospectively by a center coordinator using a tablet electronic survey. The survey will be created using a Google form questionnaire, easy to fill in and register.

The confidentiality of the patient will be protect, using patients´ identification based on their initials (first name - first last name - second last name) plus an odd or even sequential number according to the belonging hospital (ie: Mary Jo Salas Gómez MSG1).

The registry will include: demographic, cardiovascular (CV) risk factors, medical history, comorbidities, blood biochemical parameters, diagnostic imaging determinants, treatment, and outcomes data.

The information about Patient Healthe Questionnaire (PHQ) 9 questionnaire will be answered confidentially by the patient in the tablet

* Study assessment The registry consists of a descriptive cross-sectional survey. Thereby, this study is a one-time assessment, with no visit schedule
* Study limitations The main study limitation will be the failure to recruit 500 patients in the one-year period.

With respect to data limitation, the investigators will be conditioned by the information available in the medical file, and the laboratory and imaging exams requested by the head and referral physicians.

STATISTICAL METHODS Sample size and statistical power; precision assessment The sample size was estimated considering the data reported in one of the largest trials that have addressed sex differences in heart failure (HF-Action Trial by Sex, Am Heart J. 2009 Oct; 158(40): S16-S23.) 20. This trial shows that the prevalence of Heart Failure of ischemic cause (one of the main objectives of our trial) was 59% in males and 32% in females.

The calculation of the sample size was carried out to find significant differences between the prevalence of heart failure from ischemic etiology in female patients consecutively hospitalized compared to male, based on Chi-square test for comparison of proportions, considering a significance of 95% and power of 90 %. Therefore,the investigators will included in our study approximately 500 patients knowing that to get a significance of 95 % and a power of 90% the investigators must recruit at least 156 patients (52 females and 104 males) considering 2:1 male-to-female proportion. In order to perform a stratified analysis, the investigators estimated that the lowest sample size for each center should be 78 patients.( with 2:1 male -to - female proportion)

-Statistical considerations

Data management:

The data completeness and accuracy will be addressed through out-of-range alerts and control of unreported data. The nurse coordinator will verify the completeness and accuracy of the information and send the respective queries on a daily basis.

Missing data will be addressed according to covariate. Given the observational data collection of the registry, few data could be missing. These data will be addressed according the kind of covariate. In general, a multiple imputation strategy will be performed.

All the data will be electronically registered in an Excel file. Privileges will be conferred according the role of the personnel on the study. The Principal Investigators will have access to all data.

-Statistical Analyses: All the important covariates will be recorded. Specifically, information on patients' characteristics, demographics, basal functional capacity, complete blood test analyses, EKG, echocardiography, and relevant clinical information will be registered at baseline according to the protocol of each center. For analyses purposes, the prevalence of HF phenotype (ie. with preserved, mildly and reduced ejection fraction), and etiology (ie. ischemic and non ischemic) will be considered as primary outcomes.

All the variables will be tested for normality using Shapiro-Wilk test. The investigatorswill compare the percentages of heart failure with preserved ejection fraction (HFpEF), with mildly reduced ejection fraction (HFmrEF) and reduced ejection fraction (HFrEF) phenotypes according to gender, using Chi-square test. Also, the investigators will compare the percentages of HF etiology (ie. Ischemic and non ischemic) according to gender, using Chi-square test. Moreover, T-test statistics will be used according the variable.

The demographic variables that will be incorporated are:

* Age
* Sex
* Educational Level: years of education < 8, > 8 and/or < 12, >12 years
* Married, single, divorced, widowed
* Race and Ethnic origin
* Insurance status
* Family income: ≤ $ 326.000 pesos (basic income) or less U$ 500 $ 326.000 -$ 652.000 $ 652.000 - $ 1.000.000 $ 1.000.000 -$2.000.000 $ ≥ 2.000.000- <3.000.000 $ ≥ 3.000.000
* Employed, non employed, retired

The medical history that will be asked are:

* Anemia
* Smoking
* Diabetes
* Obesity
* Depression
* Hyperlipidemia
* Hypertension
* Atrial fibrillation /atrial flutter
* Ventricular arrhythmias
* Coronary disease
* Ischemic heart disease /Previous myocardial infarction (MI)
* Chronic obstructive pulmonary disease (COPD) / asthma
* Cerebrovascular disease: Ischemic Stroke /Haemorrhagic stroke / transient ischaemic attack (TIA)
* Peripheral vascular disease
* Renal insufficiency (MRDR: less 60 ml /min /m2)
* Dialysis (peritoneo/ Hemodialysis)
* Preeclampsia / Gestational Diabetes / Premature delivery
* Premature or late menarche
* Premature of late menopause
* Hyperkalemia
* Previous hospitalization
* Malignancies
* Autoimmune diseases ( i.e. Erythematosus Systemic Lupus, Rheumatoid Arthritis, Chron Disease, Vasculitis , etc)
* Genetic and Metabolic Disease (i.e. Fabry Disease, Muscular Dystrophies)

HF Characteristics.

* Preserved
* Mildly Reduced
* Reduced

HF cause: ischemic, non ischemic and hypertensive.

Decompensating HF clinical factors.

* Medication and diet non-adherence
* Atrial fibrillation /flutter
* Arrhythmias (other than AF) including bradyarrhythmias
* Infections
* Acute renal failure
* Acute coronary syndrome
* Anemia
* Pulmonary thromboembolism
* Others: specified

Precipitating clinical factors.

* Respiratory ( pneumonia and others)
* Arrhythmias
* Medication non-compliance
* Diet non-compliance
* Uncontrolled Hypertension
* Renal Failure
* Myocardial Ischemia (ACS)

Questionnaires:

* Quality of life Kansas City Cardiomyopathy Questionnaire.
* Depression: Patient Health Questionnaire 9 (PHQ-9(scale)
* HFpEF approach: The new H2FPEF (Heavy, 2 or more Hypertensive drugs, atrial Fibrillation, Pulmonary hypertension [pulmonary artery systolic pressure > 35 mmHg], Elder age > 60 years, and elevated Filling pressures [E/e´>9] ) score in patients hospitalized with HFpEF
* Frailty Score: The Frail Score

Laboratory Determinations:

* Nt-pro BNP
* Hemoglobin levels
* White blood count
* Creatinine
* Blood urea nitrogen (BUN)
* Plasma Electrolytes
* Troponin US
* Albumin
* Lipid profile
* Thyroid stimulating hormone (TSH)
* Hemoglobin A 1 C (if appropriate)
* Ferritin and Iron levels

Imaging Determinations

1. Echocardiography:

   * Ejection Fraction
   * Left Atrial volume
   * Left ventricular dimensions ( Systolic, Diastolic) and /or volumes.
   * LV segmentary motility (septal, anterior, inferior, posterior, lateral): akinesia,hypokinesia, dyskinesia( Yes/No for each one),
   * Presence of left ventricule (LV) thrombus
   * Pulmonary systolic arterial pressure
   * Mitral E/e´ratio
   * Global Longitudinal Strain
   * Valvular Regurgitations
   * Valvular Stenosis
   * Tricuspide annular plane systolic excursion (TAPSE)
2. Thoracic Radiography (RX)

   * Pulmonary congestion
   * Left Ventricular enlargement
   * Right Ventricular enlargement
   * Pleural effusion
3. Magnetic cardiac resonance

   * Late Gadolinium enhancement
   * Left ventricular volumen and ejection fraction
   * Right ventricular volumen and ejection fraction
   * Infiltrative cardiomyopathy pattern
   * Constrictive pericarditis
   * Thrombus
   * Hypertropic cardiomyopathy
4. Coronary angiogram

   * Coronary stenosis ≥ 50 %: one vessel, two vessels or three vessels
   * Coronary stenosis ≥ 70 %:
   * Coronary Occlusion
   * Ventriculography (Yes or No): ejection fraction and motility description.

Treatment

1- Pharmacological: names and daily doses

* B -blockers (total daily dose): bisoprolol, metoprolol,carvedilol, nebivolol, others
* Angiotensin converting enzyme (ACE) inhibitors (total daily dose): enalapril, ramipril, captopril, perindopril, lisinopril, others/ Angiotensin 2 Receptors blockers (total daily dose): losartan, valsartan, telmisartan, candesartan, Olmesartan, others
* Angiotensin receptor/neprilysin inhibitor (ARNI) (total daily dose): Sacubitril / Valsartan
* Mineralocorticoid antagonist receptors (total daily dose): spironolactone /eplerenone/finerenone
* Sodium glucose cotransporter 2 (SGLT 2) Inhibitors (total daily dose): dapagliflozin, empagliflozin.
* Diuretics (total daily dose): furosemide (Intravenous /oral) metolazone, hydrochlorothiazide,chlortalidone, indapamide, others
* Vericiguat
* Ivabradine
* Digoxin
* Calcium Channel Blockers: amlodipine, others
* Nitrites: Intravenous nitroglycerine/ Isosorbide dinitrate / Isosorbide mononitrate
* Other vasodilators: hydralazine
* Statins: atorvastatin, rosuvastatin, simvastatin, others
* Ezetimibe
* Anti diabetic drugs: metformin, glibenclamide, glipizide, insulin, dipeptidyl peptidase 4 (DPP4) such as sitagliptin, saxagliptin, linagliptin, vildagliptin and glucagon like peptide 1 (GLP1) analogues such as semaglutide, liraglutide, dulaglutide.
* Anticoagulants: vitamin K antagonists (VKA), direct oral anticoagulants (OACs): apixaban, rivaroxaban, dabigatran.
* Platelet inhibitors: aspirin, clopidogrel, ticagrelor.
* Intravenous Iron Therapy
* Intravenous Inotropic therapy: dobutamine, milrinone, levosimendan.

  2. Non pharmacological
* Cardiovascular Rehabilitation (Yes /No)
* Devices: Pacemaker / Cardiac resynchronization therapy/ (ICD) implantable cardioverter-defibrillator.

ELIGIBILITY:
Inclusion criteria:

* Patient with ≥ 18 years old
* Signed informed consent
* Admitted to the hospital with a :
* 1) diagnosis of acute HF as the leading cause of admission, and in which a CV therapy is needed and prescribed (ie. diuretic, vasodilator, inotropic, device), or
* 2) diagnosis of chronic HF is established during the patient hospitalization based on clinical, biochemical and/or imaging studies, and in which cardiovascular therapy is needed and prescribed (ie. diuretic, vasodilator, inotropic, device ) during the hospitalization.

Exclusion criteria:

* The patient presents a Covid 19 acute infection and/ or severe acute respiratory syndrome (SARS) -CoV 2 pneumonia is confirmed
* The patient presents a psychiatric decompensated disorder and/or a cognitive impairment which preclude assessment of this survey.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility is based on self representation of gender identity
Study Population: The study population must comply with the definition of Heart Failure according to 2021 European Society of Cardiology (ESC) Guidelines. A practical definition of HF will be shortness of breath and/or fatigue and /or ankle swelling, and/or jugular venous distention and /or rales at the lung examination, with an ejection fraction by echocardiography >= 40% ( HF with Reduced ejection fraction- HFrEF) and /or greater than 40% (41 to 49 % represents HF with midly reduced ejection fraction-HFmrEF and >= 50% Preserved Eyection Fraction-HFpEF); this last one associated with pro BNP > 125 pg/ml in sinusal rhythm.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-08-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
The prevalence of HF phenotype( preserved, mildly reduced or reduced) by sex | 12 months
  The outcome measure will be the prevalence (% of the study population) according to the HF phenotype (preserved, mildly reduced or reduced). The working definition of HF phenotypes will be in accordance to 2021 ESC guidelines of HF, based on the followimg criteria: a. clinical (shortness of breath and/or fatigue and /or ankle swelling, and/or jugular venous distention and /or rales at the lung examination),b. echocardiography: measurement of ejection fraction by transthoracic echocardiogram: HF with Reduced ejection fraction- HFrEF-(< 40%), HF with midly reduced ejection fraction-HFmrEF- (≥ 40 to 49 %) and Preserved Ejection Fraction- HFpEF- (≥ 50%), this last one associated with NT pro BNP (≥ 125 pg/ml in sinus rhythm.

SECONDARY OUTCOMES:
Prevalence of HF etiologies (ischemic, non ischemic or hypertensive) by sex. | 12 months
  The outcome measure will be the prevalence of HF etiology (ischemic, non ischemic, and hypertensive). With regard to ischemic etiology, the study definition will be based on a definite diagnosis of ischemic heart disease (epicardial coronary artery stenosis greater than 50%, and /or previous myocardial infarction, and/or previous revascularization (CABG or PCI) or a positive imaging stress test, such as echo, nuclear, or cardiac magnetic resonance (CMR) . Hypertensive cardiomyopathy will be defined for HF with reduced , mild reduced or preserved eyection fraction only if long standing hypertension (at least 20 years) , and with cardiac structural changes suitable with hypertensive etiology: presence of diastolic dysfunction, and /or LV hypertrophy.
To evaluate socioeconomic level in the study population (patients hospitalized with HF) by sex specific analysis. | 12 months
  To evaluate socioeconomic level in this cohort. The outcome measure will be based on the household average family income per capita based on the Chilean National Socioeconomic Characterization (CASEN) Survey 2020 (low from ∼276 to 340 US dollars; middle: ∼345 to 438 US dollars, and high: ∼459 to 2763 US dollars). The low socioeconomic level represents the minimum wage per capita in Chile in the study period
To evaluate educational level in the study population ( patients hospitalized with HF) by sex specific analysis. | 12 months
  To evaluate educational level in this cohort. The outcome measure will be based on the years of education.
To assess the prevalence of comorbidities associated with HF by sex-specific analysis | 12 months
  The comorbidities that will be analysed wil be: diabetes ( having a medical diagnosis of diabetes withor without pharmacological treatment or having fastingglucose ≥126 mg/dL), elderly (≥ 60 years of age, chronic renal failure (CKD) 4 or 5 phase, anemia ( hemoglobin value of less than 13.5 gm/dl in a man or less than 12.0 gm/dl in a woman), obesity (≥ 30 mg /kg 2 and Chronic obstructive pulmonary disease (COPD) based on the 2023 Global Initiative for Chronic Obstructive Lung Disease report last definition, which defines COPD as "a heterogeneous lung condition characterized by chronic respiratory symptoms (dyspnea, cough, expectoration, exacerbations) due to abnormalities of the airways (bronchitis, bronchiolitis) and/or alveoli (emphysema) that cause persistent, often progressive, airflow obstruction."
To determine the main decompensating risk factors in HF patients by sex-specific analysis | 12 months
  The prevalence of decompensating risk factors that wil be assessed will be: medication and diet non-adherence, atrial fibrillation, infections, acute renal failure and acute coronary syndromes

OTHER OUTCOMES:
To determine the presence of depressive symptoms and depression in hospitalized HF patients by a pre-specified sex analysis. | 12 months
  The outcome measure will be assessed with the Patient Health Questionnaire (PHQ)-9 , which is a validated questionnaire to measure depressive symptoms. Mild-to-moderate depressive symptoms (10 to 19 points) and major depression (≥ 20 points). The more points , the closer to the diagnosis of depression.
To determine if frailty prevalence is different in hospitalized HF patients by sex pre-specified analysis. | 12 months
  The outcome measure will be evaluated by the Simplle FRAIL questionnaire, consisting of 5 questiones. 3 or greater = frailty; 1 or 2 = prefrail

CONTACTS AND LOCATIONS:
Overall Officials: PAOLA VARLETA, MD, Principal Investigator — Fundacion de la Sociedad Chilena de Cardiologia y Cirugia Cardiovascular; MONICA ACEVEDO, MD, Principal Investigator — Fundacion de la Sociedad Chilena de Cardiologia y Cirugia Cardiovascular
Locations (1):
- Paola Varleta, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Yes
Upon request
Supporting Information: Study Protocol
Time Frame: Only available upon request to the principal investigators after the acceptance of the first publication of the study.
  For two years
Access Criteria: For international academic investigators belonging to: universities , university hospitals, public hospitals, cardiology societies , and cardiology foundations associated to cardiology colleges and associations.
URL: http://www.fundacionsochicar.cl

REFERENCES:
- [Background] McCullough PA, Philbin EF, Spertus JA, Kaatz S, Sandberg KR, Weaver WD; Resource Utilization Among Congestive Heart Failure (REACH) Study. Confirmation of a heart failure epidemic: findings from the Resource Utilization Among Congestive Heart Failure (REACH) study. J Am Coll Cardiol. 2002 Jan 2;39(1):60-9. doi: 10.1016/s0735-1097(01)01700-4. PMID 11755288
- [Background] Braunwald E. Heart failure. JACC Heart Fail. 2013 Feb;1(1):1-20. doi: 10.1016/j.jchf.2012.10.002. Epub 2013 Feb 4. PMID 24621794
- [Background] Solomon SD, Dobson J, Pocock S, Skali H, McMurray JJ, Granger CB, Yusuf S, Swedberg K, Young JB, Michelson EL, Pfeffer MA; Candesartan in Heart failure: Assessment of Reduction in Mortality and morbidity (CHARM) Investigators. Influence of nonfatal hospitalization for heart failure on subsequent mortality in patients with chronic heart failure. Circulation. 2007 Sep 25;116(13):1482-7. doi: 10.1161/CIRCULATIONAHA.107.696906. Epub 2007 Aug 27. PMID 17724259
- [Background] Diaz-Toro F, Nazzal N C, Verdejo P H. [Incidence and hospital mortality due to heart failure. Are there any differences by sex?]. Rev Med Chil. 2017 Jun;145(6):703-709. doi: 10.4067/s0034-98872017000600703. No abstract available. Spanish. PMID 29171617
- [Background] Lainscak M, Milinkovic I, Polovina M, Crespo-Leiro MG, Lund LH, Anker SD, Laroche C, Ferrari R, Coats AJS, McDonagh T, Filippatos G, Maggioni AP, Piepoli MF, Rosano GMC, Ruschitzka F, Simic D, Asanin M, Eicher JC, Yilmaz MB, Seferovic PM; European Society of Cardiology Heart Failure Long-Term Registry Investigators Group. Sex- and age-related differences in the management and outcomes of chronic heart failure: an analysis of patients from the ESC HFA EORP Heart Failure Long-Term Registry. Eur J Heart Fail. 2020 Jan;22(1):92-102. doi: 10.1002/ejhf.1645. Epub 2019 Dec 20. PMID 31863522
- [Background] Castro P, Vukasovic JL, Garces E, Sepulveda L, Ferrada M, Alvarado S; Insuficiencia Cardiaca: Registro y Organizacion. [Cardiac failure in Chilean hospitals: results of the National Registry of Heart Failure, ICARO]. Rev Med Chil. 2004 Jun;132(6):655-62. doi: 10.4067/s0034-98872004000600001. Spanish. PMID 15332366
- [Background] Vukasovic R JL, Castro G P, Sepulveda M L, Nazzal N C, Garces F E, Concepcion Ch R, Soto S JR, Yovaniniz L P, Ferrada K M, Cavada Ch G. [Characteristics of heart failure with preserved ejection fraction: results of the Chilean national registry of heart failure, ICARO]. Rev Med Chil. 2006 May;134(5):539-48. doi: 10.4067/s0034-98872006000500001. Epub 2006 Jun 19. Spanish. PMID 16802045
- [Background] Kapoor JR, Kapoor R, Ju C, Heidenreich PA, Eapen ZJ, Hernandez AF, Butler J, Yancy CW, Fonarow GC. Precipitating Clinical Factors, Heart Failure Characterization, and Outcomes in Patients Hospitalized With Heart Failure With Reduced, Borderline, and Preserved Ejection Fraction. JACC Heart Fail. 2016 Jun;4(6):464-72. doi: 10.1016/j.jchf.2016.02.017. PMID 27256749
- [Background] Jonsson A, Edner M, Alehagen U, Dahlstrom U. Heart failure registry: a valuable tool for improving the management of patients with heart failure. Eur J Heart Fail. 2010 Jan;12(1):25-31. doi: 10.1093/eurjhf/hfp175. PMID 20023041
- [Background] Adamo M, Gardner RS, McDonagh TA, Metra M. The 'Ten Commandments' of the 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2022 Feb 10;43(6):440-441. doi: 10.1093/eurheartj/ehab853. No abstract available. PMID 34922348
- [Background] Varleta P, Acevedo M, Casas-Cordero C, Berrios A, Navarrete C. Low Cardiovascular Disease Awareness in Chilean Women: Insights from the ESCI Project. Glob Heart. 2020 Aug 12;15(1):55. doi: 10.5334/gh.534. PMID 32923348
- [Background] Acevedo M, Varleta P, Casas-Cordero C, Berrios A, Navarrete C, Lopez R. Prevalence and determinants of ideal cardiovascular health in a latin women cohort: a cross-sectional study. Lancet Reg Health Am. 2021 Sep 11;4:100071. doi: 10.1016/j.lana.2021.100071. eCollection 2021 Dec. PMID 36776705
- [Background] Vogel B, Acevedo M, Appelman Y, Bairey Merz CN, Chieffo A, Figtree GA, Guerrero M, Kunadian V, Lam CSP, Maas AHEM, Mihailidou AS, Olszanecka A, Poole JE, Saldarriaga C, Saw J, Zuhlke L, Mehran R. The Lancet women and cardiovascular disease Commission: reducing the global burden by 2030. Lancet. 2021 Jun 19;397(10292):2385-2438. doi: 10.1016/S0140-6736(21)00684-X. Epub 2021 May 16. PMID 34010613
- [Background] Lichtman JH, Bigger JT Jr, Blumenthal JA, Frasure-Smith N, Kaufmann PG, Lesperance F, Mark DB, Sheps DS, Taylor CB, Froelicher ES; American Heart Association Prevention Committee of the Council on Cardiovascular Nursing; American Heart Association Council on Clinical Cardiology; American Heart Association Council on Epidemiology and Prevention; American Heart Association Interdisciplinary Council on Quality of Care and Outcomes Research; American Psychiatric Association. Depression and coronary heart disease: recommendations for screening, referral, and treatment: a science advisory from the American Heart Association Prevention Committee of the Council on Cardiovascular Nursing, Council on Clinical Cardiology, Council on Epidemiology and Prevention, and Interdisciplinary Council on Quality of Care and Outcomes Research: endorsed by the American Psychiatric Association. Circulation. 2008 Oct 21;118(17):1768-75. doi: 10.1161/CIRCULATIONAHA.108.190769. Epub 2008 Sep 29. PMID 18824640
- [Background] Bhatt KN, Kalogeropoulos AP, Dunbar SB, Butler J, Georgiopoulou VV. Depression in heart failure: Can PHQ-9 help? Int J Cardiol. 2016 Oct 15;221:246-50. doi: 10.1016/j.ijcard.2016.07.057. Epub 2016 Jul 5. PMID 27404684
- [Background] Morley JE, Vellas B, van Kan GA, Anker SD, Bauer JM, Bernabei R, Cesari M, Chumlea WC, Doehner W, Evans J, Fried LP, Guralnik JM, Katz PR, Malmstrom TK, McCarter RJ, Gutierrez Robledo LM, Rockwood K, von Haehling S, Vandewoude MF, Walston J. Frailty consensus: a call to action. J Am Med Dir Assoc. 2013 Jun;14(6):392-7. doi: 10.1016/j.jamda.2013.03.022. PMID 23764209
- [Background] Pina IL, Kokkinos P, Kao A, Bittner V, Saval M, Clare B, Goldberg L, Johnson M, Swank A, Ventura H, Moe G, Fitz-Gerald M, Ellis SJ, Vest M, Cooper L, Whellan D; HF-ACTION Investigators. Baseline differences in the HF-ACTION trial by sex. Am Heart J. 2009 Oct;158(4 Suppl):S16-23. doi: 10.1016/j.ahj.2009.07.012. PMID 19782784
- [Background] Green CP, Porter CB, Bresnahan DR, Spertus JA. Development and evaluation of the Kansas City Cardiomyopathy Questionnaire: a new health status measure for heart failure. J Am Coll Cardiol. 2000 Apr;35(5):1245-55. doi: 10.1016/s0735-1097(00)00531-3. PMID 10758967
- [Background] Reddy YNV, Carter RE, Obokata M, Redfield MM, Borlaug BA. A Simple, Evidence-Based Approach to Help Guide Diagnosis of Heart Failure With Preserved Ejection Fraction. Circulation. 2018 Aug 28;138(9):861-870. doi: 10.1161/CIRCULATIONAHA.118.034646. PMID 29792299

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/68/NCT05960968/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/68/NCT05960968/ICF_001.pdf